CLINICAL TRIAL: NCT04268966
Title: An Open-Label, Multicenter Study of the Safety and Tolerability of Brincidofovir (CMX001) for Post-Exposure Prophylaxis of Ebola Virus Disease
Brief Title: An Open-Label Study , Safety and Tolerability of Brincidofovir for Post Exposure Prophylaxis of Ebola
Acronym: BCV EBOV
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMX001-206
Record Dates: First submitted 2020-02-12; First posted 2020-02-13 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Ebola Virus Disease
MeSH Terms: conditions — Hemorrhagic Fever, Ebola | interventions — brincidofovir

ARMS (1):
- CMX001 (Experimental): Initial dose of 200mg followed by 4 doses of 100mg
  Interventions: Drug: Brincidofovir

INTERVENTIONS:
Drug: Brincidofovir
  Other Names: CMX001

SUMMARY:
The purpose of this study is to determine how safe and tolerable Brincidofovir (BCV) is when given for post exposure prophylaxis of Ebola virus disease.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and tolerability of BCV when administered for post-exposure prophylaxis of EVD

ELIGIBILITY:
Inclusion Criteria:

* Individuals have high-risk exposure to Ebola Virus based on CDC definitions
* Must be able to ingest, absorb and tolerate oral medication
* As appropriate, must be willing to use adequate methods of contraception during the study and at least 6 months after their last dose of BCV

Exclusion Criteria:

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate the safety and tolerability of BCV when administered for post-exposure prophylaxis of EVD | 8 weeks

SECONDARY OUTCOMES:
To assess the effect of BCV treatment on development of EVD in subjects through 21 days post-initiation of BCV therapy | 8 weeks